CLINICAL TRIAL: NCT00477321
Title: A Ph I/IIa Rand Placebo Ctrl, S-Blind Multictr Dose-Esc Study of SC Intermittent Interleukin-7 CYT107 in Chronically HIV-Infected Pts With CD4 T Lymphocyte Counts 101-400 Cells-/mm(3) and Plasma HIV RNA Less Than 50 Copies/mL After at Least 12 M of HAART
Brief Title: Safety Study of IL-7 in HIV-infected Patients (Inspire)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Cytheris SA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLI-107-06
Record Dates: First submitted 2007-05-22; First posted 2007-05-23 (Estimated); Last update posted 2012-10-18 (Estimated); Status verified 2012-10

CONDITIONS: HIV Infections; Lymphopenia
Keywords: Interleukin 7; Immune Reconstitution; T Cell Turnover; CD4 Lymphenia; Immune-Based Therapies; HIV Infection
MeSH Terms: conditions — HIV Infections; Lymphopenia | interventions — Interleukin-7; efineptakin alfa

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- CYT107 (Experimental): CYT107 vs Placebo (4:1 ratio)
  Interventions: Drug: CYT 107

INTERVENTIONS:
Drug: CYT 107 — 3 dose levels: 3, 10 and 20µg/kg/week.3administrations
  Other Names: CYT107; Interleukin-7; rhIL-7

SUMMARY:
This study will evaluate the safety of a new experimental drug, IL-7, in people with HIV infection. Animal studies have shown that IL-7 can improve the function and number of infection-fighting cells called T lymphocytes, or T cells. If this study shows that IL-7 is safe, additional studies will be done to see if it can improve the function or numbers of T-cells in HIV-infected persons.

HIV-infected persons who have been receiving HAART therapy for at least 12 months before enrolling in the study and have been stable on this treatment for at least 3 months before enrollment may be eligible for this study.

Participants have about 10 clinic visits over 3 months. They receive three injections of IL-7, one injection a week for 3 consecutive weeks. The injections are given as a shot under the skin in the arm or leg. On the day of each injection, the participant stays in the clinic for up to 8 hours or longer for observation and collection of blood samples. Three additional visits (one every 3 months) may be scheduled.

During the study visits the following may be done:

* Medical history, physical examination, blood tests every visit.
* Electrocardiogram (EKG) at study days 0 (day of first dose), 1, 7 (day of second dose), 14 (day of third dose) and 21.
* Chest x-ray study on day 21.
* Blood sample collections at frequent intervals during the first 96 hours after the first dose administration. A catheter (thin plastic tube) may be put into a vein in the arm and left in place to allow several blood samples to be drawn without repeated needle sticks.
* Urine tests several times during the study.

DETAILED DESCRIPTION:
Interleukin 7 (IL-7) is an essential cytokine for the thymic development and the post-thymic survival, expansion and maturation of T lymphocytes in humans. The rationale for using IL-7 as immunotherapy in HIV infection would be to support the expansion, survival and functional properties of T lymphocytes and enhance immune reconstitution. Phase I studies of a previous formulation of rhIL7 in cancer and HIV infected patients have shown that T cell proliferation and expansion can be achieved at doses that are well tolerated. The newly glycosylated form of IL-7 tested in this study has a longer half-life allowing weekly administrations.

This is a phase I/IIa, open label, single arm trial that will test the safety of three subcutaneous injections of IL-7 at three different dose levels (10, 20 and 30 micrograms/kilograms) that will be tested sequentially. Eligible subjects (400 cells/microliters greater than CD4 greater than 101 cells/microliters and VL less than 1000 copies/milliliter, on antiretroviral therapy for at least one year) will be given 3 doses of IL-7 at weekly intervals (day 0, day 7 and day 14). Participants will be followed on days 0, 1, 4, 7, 14, 21 and 28 with additional visits on days 35, 56, and 77 and optional follow up every 3 months thereafter until week 56 (approximately 1 year after enrollment). The three doses will be tested sequentially (10, 20 and 30 micrograms/kilograms per dose) and dose escalation will occur only when safety data from day 28 of the previous dose level participants are complete.

Ten subjects will enroll in each dose level and dose escalation will occur only after all subjects complete four weeks without evidence of dose-limiting toxicities. Secondary end points include a PK study of glycosylated rhIL7 as well as immunologic studies throughout the duration of the study to assess evidence of IL7 biologic activity with markers of T cell proliferation and expression of the alpha chain of the IL7 receptor. This is a multi-center international study sponsored by Cytheris with sites in USA, Canada, Italy and France. Children will be excluded and a separate study will be required in the future after the safety and biologic activity of this agent is established in adults. The study will enroll a total of approximately 30 participants.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. Age greater than or equal to 18 years
  2. HIV1 infection as documented by any licensed ELISA test kit and confirmed by Western Blot at anytime prior to study entry.
  3. On HAART for at least 12 months, and stable on treatment for at least 3 months prior to enrollment. HAART is defined as any protease inhibitor (PI or without ritonavir) + 2 nucleoside reverse transcriptase inhibitors (NNRTI) or any non nucleoside reverse transcriptase inhibitors (NNRTI) + 2 NRTIs. NOTE: RTV-boosted PIs will be considered one antiretroviral drug.
  4. CD4 cell counts greater than or equal to 101 and less than or equal to 400 cells/mm(3) on at least three consecutive measurements (including the screening value) within the previous 6 months prior to enrollment.
  5. Patient with CD4 cell counts greater than or equal to 101 and less than or equal to 150 cells/mm(3) with a NADIR greater than or equal to 50 if the NADIR was reached less than 24 months prior to enrollment.
  6. Plasma HIV RNA less than 50 copies/mL on at least two consecutive measurements (including the screening value) within the previous 6 months prior to enrollment.
  7. No AIDS-defining illness (Category C) within the last 6 months prior to enrollment
  8. Normal thyroid-stimulating hormone (TSH).
  9. Ability to understand and give written informed consent.

EXCLUSION CRITERIA:

1. Dual or single antiretroviral therapies with nucleoside analogs.
2. Enfuvirtide or any other investigational antiretroviral agent.
3. Any planned or probable modification of the antiretroviral treatment during the 3-month study period.
4. Current or recent history (less than 30 days prior to screening) of a viral, bacteria, parasitic or fungal infection requiring systemic treatment and/or hospitalization.
5. Positive PPD (North American subjects, except those who have received and completed INH prophylaxis).
6. Any serious illness requiring systemic treatment and/or hospitalization until the patient either completes therapy or is clinically stable on therapy, in the opinion of the principal investigator, for at least 28 days prior to study entry.
7. Any history of malignancy (except basal carcinoma of the skin) including any hematologic malignancy or AIDS defining malignancy, such as lymphoproliferative disorder or Kaposi's sarcoma. (Patients with Kaposi's sarcoma limited to the skin that disappeared while on HAART therapy, and without requiring any other systemic therapy, 1 year prior to study entry will be eligible to participate).
8. Any history of HIV related encephalopathy.
9. Hepatitis B or C (positive HBs Ag or positive anti HBc antibodies with a detectable HBV DNA viral load or positive anti HCV antibodies with a detectable HCV RNA viral load). Patients who became negative to HBV DNA or HCV RNA following an antiviral treatment should not be enrolled.
10. HIV-2, HTLV-1 and HTLV-2 seropositivity.
11. Pregnant or lactating women. Women of childbearing potential must have a negative serum or urine pregnancy test within 1 week prior to study entry.
12. Refusal or inability to practice contraception during therapy regardless of the gender of the patient.
13. Participation in another investigational interventional study during this study or within the last 6 months.
14. Family history of sudden cardiac death.
15. Corrected QT interval (QTc) prolongation defined as a QTc greater than or equal to 470 ms or a prior history of cardiovascular disease, arrhythmias, or significant ECG abnormalities.
16. Any history of severe auto-immune disease requiring systemic treatment or hospitalization, or any active auto-immune disease requiring treatment.
17. Any cardiac, pulmonary, thyroid, renal, hepatic, neurological (central or peripheral) disease requiring therapy and considered as significant by the investigator or a severe disorder of hemostasis.
18. Cirrhosis of any origin, and alcoholic or non alcoholic steatohepatitis, either proven histologically or only suspected.
19. Any gastrointestinal illness associated with chronic or intermittent diarrhea.
20. Hypertension with a resting systolic blood pressure greater than 140 mmHg or a resting diastolic blood pressure greater than 90 mmHg despite adequate antihypertensive treatment.
21. Use of tipranavir/ritonavir (TPV/r).
22. Previous treatment with IL-2 or IL-7 at any time prior to study entry.
23. Prior treatment with immunomodulatory agents such as growth factors, immunosuppressive drugs, cytotoxic chemotherapy or hydroxyurea within 3 months of study entry.
24. Use of systemic corticosteroids within 3 months prior to enrollment.
25. Any vaccination within 30 days prior to study entry and during the study (until follow-up at W12).
26. Need for anticoagulant medication.
27. History of splenectomy.
28. Any hematologic disease associated with hypersplenism, such as thalassemia, hereditary spherocytosis, Gaucher's disease, and autoimmune haemolytic anemia.
29. Nephrological abnormalities: Calculated creatinine clearance less than 90 ml/min (according to Cockroft formula) or proteinuria greater than 300 mg/l.
30. Other abnormal laboratory findings: hemaglobin less than 10g/dl; Neutrophils less than 1,000/mm(3); Platelets less than 100,000/mm(3); AST, ALT, or Alk. Phosph. greater than 2.5 x ULN; Total bilirubin greater than 1.5 x ULN (or greater than 5 x ULN if the patient is treated by atazanavir or by indinavir, and if the increase is due to unconjugated bilirubin and if liver enzymes are normal); Lipase greater than 2 x ULN; PT/PPT greater than 1.5 x ULN.
31. Poor compliance on HAART or any other chronic treatment in the opinion of the investigator.
32. Active drug or alcohol use or dependence that, in the opinion of the investigator, would interfere with adherence to study requirements. Patients must agree to refrain from substance abuse use during the course of the study.
33. Any past or current psychiatric illness that, in the opinion of the investigator, would interfere with adherence to study requirements or the ability and willingness to give written informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2007-05; Primary Completion 2009-10 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Safety | 12 weeks

SECONDARY OUTCOMES:
Changes in T cell counts, changes in T cell proliferation, changes in expression of CD127 on T cells | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Michael Lederman, Study Chair — Case Western Reserve University; Yves Levy, Study Chair — Hopital Henri Mondor; Irini Sereti, Study Chair — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (8):
- United States (3):
  - University of Miami School of Medicine, Miami, Florida
  - National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland
  - Case Western Reserve University, Cleveland, Ohio
- McGill University Health Center (MUHC), Montreal, Canada
- France (3):
  - Hopital Henri Mendor-Service d'Immunologie Clinique, Créteil
  - Hopital Kremlin Bicêtre, Le Kremlin-Bicêtre
  - Hopital Saint Louis, Paris
- San Raffaele Scientific Institute, Milan, Italy

REFERENCES:
- [Background] Stebbing J, Gazzard B, Douek DC. Where does HIV live? N Engl J Med. 2004 Apr 29;350(18):1872-80. doi: 10.1056/NEJMra032395. No abstract available. PMID 15115833
- [Background] Battegay M, Nuesch R, Hirschel B, Kaufmann GR. Immunological recovery and antiretroviral therapy in HIV-1 infection. Lancet Infect Dis. 2006 May;6(5):280-7. doi: 10.1016/S1473-3099(06)70463-7. PMID 16631548
- [Background] Douek DC, Picker LJ, Koup RA. T cell dynamics in HIV-1 infection. Annu Rev Immunol. 2003;21:265-304. doi: 10.1146/annurev.immunol.21.120601.141053. Epub 2001 Dec 19. PMID 12524385
- See also: NIH Clinical Center Detailed Web Page — http://clinicalstudies.info.nih.gov/detail/A_2007-I-0155.html